CLINICAL TRIAL: NCT04538833
Title: Monosialoganglioside in the Treatment of Neurotoxicity Induced by Albumin-bound Paclitaxel : a Multicenter, Double-blind, Randomized Controlled Phase II Clinical Trial
Brief Title: GM1 in the Treatment of Neurotoxicity Induced by Albumin-bound Paclitaxel
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: In the clinical treatment, no patient with a score of less than 38(FACT Ntx Score) points after 1-2 weeks of application of albumin bound paclitaxel in this project, therefore, there is no suitable subject after screening
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Zhenzhen Liu, Director, Henan Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HNCH-BC007
Record Dates: First submitted 2020-08-30; First posted 2020-09-04 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Early Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- monosialic ganglioside (Experimental): On the days -1, 1, and 2 of albumin-bound paclitaxel application, 80 mg of monosialic ganglioside were applied (monosialic ganglioside was a single infusion)
  Interventions: Drug: monosialic gangliosides
- Placebo (Placebo Comparator): The control group received placebo on days -1, 1, and 2 of albumin-bound paclitaxel application, (placebo as a single infusion)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: monosialic gangliosides — The experimental group received 80 mg of monosialic gangliosides (GM1) on days -1, 1, and 2 of albumin-bound paclitaxel(GM1 is a single infusion).
  Arms: monosialic ganglioside
Other: Placebo — The control group received placebo on days -1, 1, and 2 of albumin-bound paclitaxel (placebo as a single infusion)
  Arms: Placebo

SUMMARY:
Taxane-induced peripheral neuropathy (TIPN) caused by albumin-bound paclitaxel is a dose-limiting toxicity. The main symptoms of discomfort are numbness, tingling, and burning sensations in the glove-sock-like distribution of the limbs. At present, there are few effective methods for clinical treatment of TIPN, and there is no widely agreed consensus on effective treatment in the world. Therefore, it is of great clinical significance and practical value to carry out clinical research to explore drugs to relieve TIPN.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients diagnosed with early breast cancer by histology;
2. Age ≥18 years old and ≤75 years old
3. At least 1-2 cycles of standard chemotherapy regimens containing albumin-bound paclitaxel were used in adjuvant / neoadjuvant chemotherapy regimens, The FACT-Ntx score was ≤ 37, and the remaining chemotherapy cycles were at least 2 cycles. the standard regimen included: a, albumin paclitaxel one-week regimen; b, albumin paclitaxel 3-week regimen. Platinum and other types of neurotoxic drugs shall not be included in the regimen.
4. ECOG score of the patient is ≤1;
5. Expected survival time ≥ 3 months;
6. The function level of main organs must meet the following requirements (no blood transfusion and no use of leukocyte or platelet rising drugs within 2 weeks before screening) Blood routine: neutrophil (ANC) ≥ 1.5x 10^9 / L; platelet (PLT) ≥ 90x10^9 / L; hemoglobin (Hb) ≥ 90g / L; Blood biochemical total bilirubin (TBIL) ≤ 1.5xULN; alanine aminotransferase (AST) and aspartate aminotransferase (AST) not exceeding 2×ULN; blood urea nitrogen (BUN) and creatinine (CR) below 1.5 × ULN;
7. FACT-Ntx score is 44 points before the adjuvant / neoadjuvant chemotherapy was given;
8. Sign the informed consent.

Exclusion Criteria:

1. Other pathological symptoms or diseases may affect the assessment of adverse neurotoxicity before enrollment
2. Patients receiving other medications may cause similar adverse neurotoxic effects within 4 weeks before treatment with this regimen, or they may also receive neurotoxic medications at the same time. Including paclitaxel or analogues; vinca alkaloids or analogues; platinums or analogues; cytarabine, thalidomide, bortezomib or cabazine; other drugs or treatments may cause peripheral neurotoxicity;
3. Patients with poor overall condition and ECOG score> 1;
4. pregnant or lactating women;
5. Patients who also suffer from other neurological abnormalities cannot accurately record the occurrence and severity of neurotoxicity;
6. The patient is known to be allergic to the test drug or excipient ingredients of these products;
7. Patients with hereditary abnormalities of glucose and lipid metabolism (gangliopathies, such as idiopathic and retinopathy of triad families);
8. Patients not suitable for ganglioside treatment;
9. Patients with severe concurrent diseases may endanger safety and interfere with scheduled treatment, or the combination of diseases may affect the completion of the study, depending on the judgment of the investigator.
10. Patients with a clear history of neurological or mental disorders, including epilepsy or dementia.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2022-08-22 (Actual)

PRIMARY OUTCOMES:
FACT-Ntx score | 2 weeks after chemotherapy
  The FACT-Ntx subscale includes 11 items, each of which is divided into 5 scoring levels: 0, 1, 2, 3, 4, and a total score of 44. Higher scores indicate lower side effects

SECONDARY OUTCOMES:
CTCAE Version 4.0 score | During chemotherapy, and 2 weeks, 3 months, 6 months, and 12 months after chemotherapy
  Peripheral sensory neuropathy, peripheral motor neuropathy, paresthesia, myalgia, arthralgia, and neuralgia were evaluated by the CTCAE 4.0 rating scale. Each item was divided into 5 levels: 1, 2, 3, 4, 5, Higher indicates higher neurotoxicity
FACT-Taxane score | During chemotherapy, and 2 weeks, 3 months, 6 months, and 12 months after chemotherapy
  The FACT-Taxane scale contains 16 items, each item is divided into 5 grades: 0, 1, 2, 3, 4, with a total score of 64. The higher the score, the lower the side effects.
FACT-G score | During chemotherapy, and 2 weeks, 3 months, 6 months, and 12 months after chemotherapy
  The FACT-G Scale contains 27 items, each item is divided into 5 grades: 0, 1, 2, 3, 4, with a total score of 108
FACT-Ntx score | 3 months, 6 months, and 12 months after chemotherapy
  The FACT-Ntx subscale includes 11 items, each of which is divided into 5 scoring levels: 0, 1, 2, 3, 4, and a total score of 44. Higher scores indicate lower side effects

CONTACTS AND LOCATIONS:
Overall Officials: Zhenzhen Liu, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China